CLINICAL TRIAL: NCT01006135
Title: Spiriva Observational Study Measuring Saint George's Respiratory Questionnaire (SGRQ) in Routine Medical Practice in Central & Eastern European Region
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.450
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- COPD patients

SUMMARY:
The objective of this observational study is to collect and evaluate data on Health Related Quality of Life (HRQoL) of Spiriva delivered by HandiHaler, using disease specific SGRQ in the national samples of Central & Central European patients with varying severities of chronic obstructive pulmonary disease (COPD) in the real life setting over the 6 months.

DETAILED DESCRIPTION:
Study Design:

an open-label, uncontrolled and single arm post-marketing surveillance study

ELIGIBILITY:
Inclusion criteria:

* 40 years and older male and female ambulatory outpatients.
* Clinical diagnosis of Chronic Obstructive Lung Disease (COPD) (Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines: Forced expiratory Volume in one second (FEV1)/ Forced Vital Capacity (FVC) < 0.7 and FEV1 < 80% predicted).
* Stable patient, without exacerbation for at least one month to the study.

Exclusion criteria:

* Uncooperative patients as judged by the physician.
* Patients that have any condition which, according to the participating physician's opinion, might decrease the chance of obtaining satisfactory data to achieve the objectives of the observation study.
* Patients with any conditions excluded as per Country specific package insert.
* Patients currently enrolled in another clinical trial which requires a change in medication for their respiratory problems.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 4852 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (864):
- Croatia (22):
  - Boehringer Ingelheim Investigational Site 1, Drniš
  - Boehringer Ingelheim Investigational Site 2, Ivani? Grad-Zagreb
  - Boehringer Ingelheim Investigational Site 3, Karlovac
  - Boehringer Ingelheim Investigational Site 4, Knin
  - Boehringer Ingelheim Investigational Site 5, Metkovi?
  - Boehringer Ingelheim Investigational Site 6, Osijek
  - Boehringer Ingelheim Investigational Site 7, Osijek
  - Boehringer Ingelheim Investigational Site 8, Petrinja-Sisak
  - Boehringer Ingelheim Investigational Site 9, Požega
  - Boehringer Ingelheim Investigational Site 10, Pula
  - Boehringer Ingelheim Investigational Site 11, Rijeka
  - Boehringer Ingelheim Investigational Site 12, Rijeka
  - Boehringer Ingelheim Investigational Site 13, Samobor
  - Boehringer Ingelheim Investigational Site 14, Senj
  - Boehringer Ingelheim Investigational Site 16, Slavonski Brod
  - Boehringer Ingelheim Investigational Site 15, Šibenik
  - Boehringer Ingelheim Investigational Site 17, Vinkovci
  - Boehringer Ingelheim Investigational Site 18, Virovitica
  - Boehringer Ingelheim Investigational Site 19, Vukovar
  - Boehringer Ingelheim Investigational Site 20, Zadar
  - Boehringer Ingelheim Investigational Site 21, Zagreb
  - Boehringer Ingelheim Investigational Site 22, Zagreb
- Poland (438):
  - Boehringer Ingelheim Investigational Site 23, Aleksandrów Kujawski
  - Boehringer Ingelheim Investigational Site 24, Augustów
  - Boehringer Ingelheim Investigational Site 25, Belsk Duży
  - Boehringer Ingelheim Investigational Site 27, Bialystok
  - Boehringer Ingelheim Investigational Site 28, Bialystok
  - Boehringer Ingelheim Investigational Site 29, Bialystok
  - Boehringer Ingelheim Investigational Site 30, Bialystok
  - Boehringer Ingelheim Investigational Site 31, Bialystok
  - Boehringer Ingelheim Investigational Site 32, Bialystok
  - Boehringer Ingelheim Investigational Site 33, Bialystok
  - Boehringer Ingelheim Investigational Site 34, Bialystok
  - Boehringer Ingelheim Investigational Site 26, Biała Prudnicka
  - Boehringer Ingelheim Investigational Site 35, Bielawa
  - Boehringer Ingelheim Investigational Site 36, Bielawa
  - Boehringer Ingelheim Investigational Site 37, Bielsk
  - Boehringer Ingelheim Investigational Site 38, Bielsko-Biala
  - Boehringer Ingelheim Investigational Site 39, Biskupcu
  - Boehringer Ingelheim Investigational Site 40, Bochnia
  - Boehringer Ingelheim Investigational Site 41, Bolesław
  - Boehringer Ingelheim Investigational Site 42, Bolesławiec
  - Boehringer Ingelheim Investigational Site 43, Brodnica
  - Boehringer Ingelheim Investigational Site 44, Brzesko
  - Boehringer Ingelheim Investigational Site 45, Brzeziny
  - Boehringer Ingelheim Investigational Site 46, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 47, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 48, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 49, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 50, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 51, Bystra
  - Boehringer Ingelheim Investigational Site 52, Bystra
  - Boehringer Ingelheim Investigational Site 53, Bytom
  - Boehringer Ingelheim Investigational Site 54, Bytom
  - Boehringer Ingelheim Investigational Site 55, Cewice
  - Boehringer Ingelheim Investigational Site 57, Chełm
  - Boehringer Ingelheim Investigational Site 58, Chełmno
  - Boehringer Ingelheim Investigational Site 59, Chełmża
  - Boehringer Ingelheim Investigational Site 56, Chęciny
  - Boehringer Ingelheim Investigational Site 60, Chodzież
  - Boehringer Ingelheim Investigational Site 61, Chojnice
  - Boehringer Ingelheim Investigational Site 62, Chorzów
  - Boehringer Ingelheim Investigational Site 63, Chorzów
  - Boehringer Ingelheim Investigational Site 64, Chorzów
  - Boehringer Ingelheim Investigational Site 65, Chrzanów
  - Boehringer Ingelheim Investigational Site 66, Ciechanów
  - Boehringer Ingelheim Investigational Site 67, Ciechanów
  - Boehringer Ingelheim Investigational Site 68, Cieszyn
  - Boehringer Ingelheim Investigational Site 69, Czechowice-Dziedzice
  - Boehringer Ingelheim Investigational Site 70, Czerwin
  - Boehringer Ingelheim Investigational Site 71, Częstochowa
  - Boehringer Ingelheim Investigational Site 72, Częstochowa
  - Boehringer Ingelheim Investigational Site 73, Częstochowa
  - Boehringer Ingelheim Investigational Site 74, Czluchów
  - Boehringer Ingelheim Investigational Site 75, Dabrowa Górnicza
  - Boehringer Ingelheim Investigational Site 76, Dabrowa Górnicza
  - Boehringer Ingelheim Investigational Site 77, Dabrowa Górnicza
  - Boehringer Ingelheim Investigational Site 78, Dabrowa Niemodlinska
  - Boehringer Ingelheim Investigational Site 79, Dobrzechów
  - Boehringer Ingelheim Investigational Site 80, Dobrzeń Wielki
  - Boehringer Ingelheim Investigational Site 81, Dziergowice
  - Boehringer Ingelheim Investigational Site 82, Dzierzenin
  - Boehringer Ingelheim Investigational Site 83, Elblag
  - Boehringer Ingelheim Investigational Site 84, Elblag
  - Boehringer Ingelheim Investigational Site 85, Elblag
  - Boehringer Ingelheim Investigational Site 86, Ełk
  - Boehringer Ingelheim Investigational Site 87, Garwolin
  - Boehringer Ingelheim Investigational Site 88, Garwolin
  - Boehringer Ingelheim Investigational Site 89, Gdansk
  - Boehringer Ingelheim Investigational Site 90, Gdansk
  - Boehringer Ingelheim Investigational Site 91, Gdansk
  - Boehringer Ingelheim Investigational Site 92, Gdansk
  - Boehringer Ingelheim Investigational Site 93, Gdansk
  - Boehringer Ingelheim Investigational Site 94, Gdansk
  - Boehringer Ingelheim Investigational Site 95, Gdynia
  - Boehringer Ingelheim Investigational Site 96, Gdynia
  - Boehringer Ingelheim Investigational Site 97, Gierałtowice
  - Boehringer Ingelheim Investigational Site 98, Giżycko
  - Boehringer Ingelheim Investigational Site 100, Gliwice
  - Boehringer Ingelheim Investigational Site 101, Gliwice
  - Boehringer Ingelheim Investigational Site 99, Gliwice
  - Boehringer Ingelheim Investigational Site 102, Glogów
  - Boehringer Ingelheim Investigational Site 103, Glogów
  - Boehringer Ingelheim Investigational Site 104, Glogów
  - Boehringer Ingelheim Investigational Site 160, Gmina Koszęcin
  - Boehringer Ingelheim Investigational Site 270, Gmina Poddębice
  - Boehringer Ingelheim Investigational Site 334, Gmina Śrem
  - Boehringer Ingelheim Investigational Site 352, Gmina Świecie
  - Boehringer Ingelheim Investigational Site 375, Gmina Uchanie
  - Boehringer Ingelheim Investigational Site 107, Gniezno
  - Boehringer Ingelheim Investigational Site 108, Gniezno
  - Boehringer Ingelheim Investigational Site 109, Golub-Dobrzyń
  - Boehringer Ingelheim Investigational Site 110, Gorlice
  - Boehringer Ingelheim Investigational Site 112, Gorzów Wlkp
  - Boehringer Ingelheim Investigational Site 113, Gorzów Wlkp
  - Boehringer Ingelheim Investigational Site 111, Górno
  - Boehringer Ingelheim Investigational Site 114, Grodzisk Mazowiecki
  - Boehringer Ingelheim Investigational Site 115, Grodzisk Mazowiecki
  - Boehringer Ingelheim Investigational Site 116, Grodzisk Wielkopolski
  - Boehringer Ingelheim Investigational Site 117, Grójec
  - Boehringer Ingelheim Investigational Site 118, Grudziądz
  - Boehringer Ingelheim Investigational Site 119, Grudziądz
  - Boehringer Ingelheim Investigational Site 120, Gryfice
  - Boehringer Ingelheim Investigational Site 105, Głuchołazy
  - Boehringer Ingelheim Investigational Site 106, Głuchołazy
  - Boehringer Ingelheim Investigational Site 121, Hajnówka
  - Boehringer Ingelheim Investigational Site 122, Hrubieszów
  - Boehringer Ingelheim Investigational Site 124, Inowrocław
  - Boehringer Ingelheim Investigational Site 125, Inowrocław
  - Boehringer Ingelheim Investigational Site 126, Inowrocław
  - Boehringer Ingelheim Investigational Site 123, Iława
  - Boehringer Ingelheim Investigational Site 128, Jaroszowiec
  - Boehringer Ingelheim Investigational Site 127, Jarosław
  - Boehringer Ingelheim Investigational Site 132, Jastrzębie Zdrój
  - Boehringer Ingelheim Investigational Site 133, Jastrzębie Zdrój
  - Boehringer Ingelheim Investigational Site 129, Jasło
  - Boehringer Ingelheim Investigational Site 130, Jasło
  - Boehringer Ingelheim Investigational Site 131, Jasło
  - Boehringer Ingelheim Investigational Site 134, Jaworzno
  - Boehringer Ingelheim Investigational Site 135, Jejkowice
  - Boehringer Ingelheim Investigational Site 136, Kalej
  - Boehringer Ingelheim Investigational Site 137, Katowice
  - Boehringer Ingelheim Investigational Site 138, Katowice
  - Boehringer Ingelheim Investigational Site 139, Katowice
  - Boehringer Ingelheim Investigational Site 140, Katowice
  - Boehringer Ingelheim Investigational Site 141, Katowice
  - Boehringer Ingelheim Investigational Site 142, Katowice
  - Boehringer Ingelheim Investigational Site 143, Katowice
  - Boehringer Ingelheim Investigational Site 144, Katowice
  - Boehringer Ingelheim Investigational Site 145, Kędzierzyn-Koźle
  - Boehringer Ingelheim Investigational Site 146, Kępno
  - Boehringer Ingelheim Investigational Site 147, Kielce
  - Boehringer Ingelheim Investigational Site 148, Kielce
  - Boehringer Ingelheim Investigational Site 149, Kielce
  - Boehringer Ingelheim Investigational Site 155, Komorniki
  - Boehringer Ingelheim Investigational Site 156, Konin
  - Boehringer Ingelheim Investigational Site 157, Konin
  - Boehringer Ingelheim Investigational Site 159, Koszalin
  - Boehringer Ingelheim Investigational Site 161, Kowary
  - Boehringer Ingelheim Investigational Site 162, Kozienice
  - Boehringer Ingelheim Investigational Site 154, Kołobrzeg
  - Boehringer Ingelheim Investigational Site 158, Kórnik
  - Boehringer Ingelheim Investigational Site 163, Krakow
  - Boehringer Ingelheim Investigational Site 164, Krakow
  - Boehringer Ingelheim Investigational Site 165, Krakow
  - Boehringer Ingelheim Investigational Site 166, Krakow
  - Boehringer Ingelheim Investigational Site 167, Krakow
  - Boehringer Ingelheim Investigational Site 168, Krakow
  - Boehringer Ingelheim Investigational Site 169, Krakow
  - Boehringer Ingelheim Investigational Site 170, Krakow
  - Boehringer Ingelheim Investigational Site 171, Krakow
  - Boehringer Ingelheim Investigational Site 172, Krakow
  - Boehringer Ingelheim Investigational Site 173, Krakow
  - Boehringer Ingelheim Investigational Site 174, Krakow
  - Boehringer Ingelheim Investigational Site 175, Kraśnik
  - Boehringer Ingelheim Investigational Site 176, Krosno
  - Boehringer Ingelheim Investigational Site 177, Krosno
  - Boehringer Ingelheim Investigational Site 178, Krzeszowice
  - Boehringer Ingelheim Investigational Site 179, Kutno
  - Boehringer Ingelheim Investigational Site 150, Kłodawa
  - Boehringer Ingelheim Investigational Site 151, Kłodawa
  - Boehringer Ingelheim Investigational Site 152, Kłodzko
  - Boehringer Ingelheim Investigational Site 153, Kłodzko
  - Boehringer Ingelheim Investigational Site 183, Legionowo
  - Boehringer Ingelheim Investigational Site 184, Legionowo
  - Boehringer Ingelheim Investigational Site 185, Legnica
  - Boehringer Ingelheim Investigational Site 181, Lębork
  - Boehringer Ingelheim Investigational Site 182, Lębork
  - Boehringer Ingelheim Investigational Site 186, Lipsko
  - Boehringer Ingelheim Investigational Site 202, Lowicz
  - Boehringer Ingelheim Investigational Site 187, Lódz
  - Boehringer Ingelheim Investigational Site 188, Lódz
  - Boehringer Ingelheim Investigational Site 189, Lódz
  - Boehringer Ingelheim Investigational Site 190, Lódz
  - Boehringer Ingelheim Investigational Site 191, Lódz
  - Boehringer Ingelheim Investigational Site 192, Lódz
  - Boehringer Ingelheim Investigational Site 193, Lódz
  - Boehringer Ingelheim Investigational Site 194, Lódz
  - Boehringer Ingelheim Investigational Site 195, Lódz
  - Boehringer Ingelheim Investigational Site 196, Lódz
  - Boehringer Ingelheim Investigational Site 197, Lódz
  - Boehringer Ingelheim Investigational Site 198, Lódz
  - Boehringer Ingelheim Investigational Site 199, Lódz
  - Boehringer Ingelheim Investigational Site 200, Lódz
  - Boehringer Ingelheim Investigational Site 203, Lubin
  - Boehringer Ingelheim Investigational Site 204, Lubin
  - Boehringer Ingelheim Investigational Site 205, Lubin
  - Boehringer Ingelheim Investigational Site 206, Lublin
  - Boehringer Ingelheim Investigational Site 207, Lubliniec
  - Boehringer Ingelheim Investigational Site 208, Lubomierz
  - Boehringer Ingelheim Investigational Site 209, Makow Maz
  - Boehringer Ingelheim Investigational Site 210, Malanów
  - Boehringer Ingelheim Investigational Site 211, Malbork
  - Boehringer Ingelheim Investigational Site 213, Marki
  - Boehringer Ingelheim Investigational Site 212, Małdyty
  - Boehringer Ingelheim Investigational Site 214, Miechów
  - Boehringer Ingelheim Investigational Site 216, Mielec
  - Boehringer Ingelheim Investigational Site 217, Mielec
  - Boehringer Ingelheim Investigational Site 215, Międzyrzecz
  - Boehringer Ingelheim Investigational Site 218, Morąg
  - Boehringer Ingelheim Investigational Site 221, Myszków
  - Boehringer Ingelheim Investigational Site 220, Mysłowice
  - Boehringer Ingelheim Investigational Site 219, Myślenice
  - Boehringer Ingelheim Investigational Site 222, Nasielsk
  - Boehringer Ingelheim Investigational Site 223, Nisko
  - Boehringer Ingelheim Investigational Site 224, Niwiski
  - Boehringer Ingelheim Investigational Site 225, Nowa Dęba
  - Boehringer Ingelheim Investigational Site 226, Nowa Dęba
  - Boehringer Ingelheim Investigational Site 227, Nowy Dwór Maz
  - Boehringer Ingelheim Investigational Site 228, Nowy Sącz
  - Boehringer Ingelheim Investigational Site 229, Nowy Sącz
  - Boehringer Ingelheim Investigational Site 230, Nowy Sącz
  - Boehringer Ingelheim Investigational Site 231, Nowy Sącz
  - Boehringer Ingelheim Investigational Site 232, Nowy Tomyśl
  - Boehringer Ingelheim Investigational Site 233, Oborniki
  - Boehringer Ingelheim Investigational Site 240, Olesno
  - Boehringer Ingelheim Investigational Site 241, Olesno
  - Boehringer Ingelheim Investigational Site 237, Oleśnica
  - Boehringer Ingelheim Investigational Site 238, Oleśnica
  - Boehringer Ingelheim Investigational Site 239, Oleśnica
  - Boehringer Ingelheim Investigational Site 242, Olkusz
  - Boehringer Ingelheim Investigational Site 243, Olsztyn
  - Boehringer Ingelheim Investigational Site 244, Olsztyn
  - Boehringer Ingelheim Investigational Site 245, Olsztyn
  - Boehringer Ingelheim Investigational Site 246, Opatów
  - Boehringer Ingelheim Investigational Site 247, Opoczno
  - Boehringer Ingelheim Investigational Site 248, Opole
  - Boehringer Ingelheim Investigational Site 249, Opole
  - Boehringer Ingelheim Investigational Site 250, Opole
  - Boehringer Ingelheim Investigational Site 251, Opole
  - Boehringer Ingelheim Investigational Site 252, Opole
  - Boehringer Ingelheim Investigational Site 253, Orzese
  - Boehringer Ingelheim Investigational Site 254, Ostrowiec/Sandomierz
  - Boehringer Ingelheim Investigational Site 255, Oświęcim
  - Boehringer Ingelheim Investigational Site 256, Otwock
  - Boehringer Ingelheim Investigational Site 257, Otwock
  - Boehringer Ingelheim Investigational Site 258, Otwock
  - Boehringer Ingelheim Investigational Site 234, Oława
  - Boehringer Ingelheim Investigational Site 235, Oława
  - Boehringer Ingelheim Investigational Site 236, Oława
  - Boehringer Ingelheim Investigational Site 259, Pabianice
  - Boehringer Ingelheim Investigational Site 260, Pabianice
  - Boehringer Ingelheim Investigational Site 261, Pajęczno
  - Boehringer Ingelheim Investigational Site 264, Pinczów
  - Boehringer Ingelheim Investigational Site 265, Piotrkow Tybunalski
  - Boehringer Ingelheim Investigational Site 262, Piła
  - Boehringer Ingelheim Investigational Site 263, Piła
  - Boehringer Ingelheim Investigational Site 266, Pleszew
  - Boehringer Ingelheim Investigational Site 271, Polanica-Zdrój
  - Boehringer Ingelheim Investigational Site 272, Poznan
  - Boehringer Ingelheim Investigational Site 273, Poznan
  - Boehringer Ingelheim Investigational Site 274, Poznan
  - Boehringer Ingelheim Investigational Site 275, Poznan
  - Boehringer Ingelheim Investigational Site 276, Poznan
  - Boehringer Ingelheim Investigational Site 277, Poznan
  - Boehringer Ingelheim Investigational Site 278, Poznan
  - Boehringer Ingelheim Investigational Site 279, Poznan
  - Boehringer Ingelheim Investigational Site 280, Poznan
  - Boehringer Ingelheim Investigational Site 281, Poznan
  - Boehringer Ingelheim Investigational Site 282, Poznan
  - Boehringer Ingelheim Investigational Site 283, Prabuty
  - Boehringer Ingelheim Investigational Site 284, Proszowice
  - Boehringer Ingelheim Investigational Site 285, Proszowice
  - Boehringer Ingelheim Investigational Site 286, Proszowice
  - Boehringer Ingelheim Investigational Site 287, Przemyśl
  - Boehringer Ingelheim Investigational Site 288, Przemyśl
  - Boehringer Ingelheim Investigational Site 289, Pszczyna
  - Boehringer Ingelheim Investigational Site 290, Puck
  - Boehringer Ingelheim Investigational Site 291, Puławy
  - Boehringer Ingelheim Investigational Site 267, Płock
  - Boehringer Ingelheim Investigational Site 268, Płock
  - Boehringer Ingelheim Investigational Site 269, Płock
  - Boehringer Ingelheim Investigational Site 292, Racibórz
  - Boehringer Ingelheim Investigational Site 293, Racibórz
  - Boehringer Ingelheim Investigational Site 294, Radlin
  - Boehringer Ingelheim Investigational Site 295, Radom
  - Boehringer Ingelheim Investigational Site 296, Radom
  - Boehringer Ingelheim Investigational Site 297, Radom
  - Boehringer Ingelheim Investigational Site 298, Radomsko
  - Boehringer Ingelheim Investigational Site 299, Radomsko
  - Boehringer Ingelheim Investigational Site 300, Radomsko
  - Boehringer Ingelheim Investigational Site 301, Radziejów
  - Boehringer Ingelheim Investigational Site 302, Rawa Mazowiecka
  - Boehringer Ingelheim Investigational Site 303, Rawicz
  - Boehringer Ingelheim Investigational Site 304, Rawicz
  - Boehringer Ingelheim Investigational Site 305, Reda
  - Boehringer Ingelheim Investigational Site 306, Rodzinna
  - Boehringer Ingelheim Investigational Site 307, Rokitno
  - Boehringer Ingelheim Investigational Site 308, Ruda Śląska
  - Boehringer Ingelheim Investigational Site 309, Rumia
  - Boehringer Ingelheim Investigational Site 310, Rybnik
  - Boehringer Ingelheim Investigational Site 311, Rypin
  - Boehringer Ingelheim Investigational Site 312, Rzeszów
  - Boehringer Ingelheim Investigational Site 313, Rzeszów
  - Boehringer Ingelheim Investigational Site 314, Sanok
  - Boehringer Ingelheim Investigational Site 315, Sejny
  - Boehringer Ingelheim Investigational Site 316, Siedlce
  - Boehringer Ingelheim Investigational Site 317, Siemianowice Śląskie
  - Boehringer Ingelheim Investigational Site 318, Sieradz
  - Boehringer Ingelheim Investigational Site 320, Skawina
  - Boehringer Ingelheim Investigational Site 319, Skąpe
  - Boehringer Ingelheim Investigational Site 321, Skwierzyna
  - Boehringer Ingelheim Investigational Site 324, Sobków
  - Boehringer Ingelheim Investigational Site 325, Sochaczew
  - Boehringer Ingelheim Investigational Site 326, Sochaczew
  - Boehringer Ingelheim Investigational Site 327, Sokolów Podlaski
  - Boehringer Ingelheim Investigational Site 328, Sopot
  - Boehringer Ingelheim Investigational Site 329, Sosnowiec
  - Boehringer Ingelheim Investigational Site 330, Sosnowiec
  - Boehringer Ingelheim Investigational Site 331, Sosnowiec
  - Boehringer Ingelheim Investigational Site 332, Sosnowiec
  - Boehringer Ingelheim Investigational Site 333, Sosnowiec
  - Boehringer Ingelheim Investigational Site 336, Stalowa Wola
  - Boehringer Ingelheim Investigational Site 337, Starachowice
  - Boehringer Ingelheim Investigational Site 338, Stare Miasto
  - Boehringer Ingelheim Investigational Site 339, Stargard
  - Boehringer Ingelheim Investigational Site 340, Stargard
  - Boehringer Ingelheim Investigational Site 341, Starogard Gdański
  - Boehringer Ingelheim Investigational Site 342, Starogard Gdański
  - Boehringer Ingelheim Investigational Site 343, Staroźreby
  - Boehringer Ingelheim Investigational Site 344, Staszów
  - Boehringer Ingelheim Investigational Site 345, Stryków
  - Boehringer Ingelheim Investigational Site 346, Strzegom
  - Boehringer Ingelheim Investigational Site 347, Strzyzów
  - Boehringer Ingelheim Investigational Site 348, Sulisławice
  - Boehringer Ingelheim Investigational Site 349, Suwałki
  - Boehringer Ingelheim Investigational Site 350, Suwałki
  - Boehringer Ingelheim Investigational Site 351, Swarzędz
  - Boehringer Ingelheim Investigational Site 354, Szczecin
  - Boehringer Ingelheim Investigational Site 355, Szczecin
  - Boehringer Ingelheim Investigational Site 356, Szczecin
  - Boehringer Ingelheim Investigational Site 357, Szczytno
  - Boehringer Ingelheim Investigational Site 358, Sztum
  - Boehringer Ingelheim Investigational Site 322, Słupca
  - Boehringer Ingelheim Investigational Site 323, Słupsk
  - Boehringer Ingelheim Investigational Site 335, Środa Śląska
  - Boehringer Ingelheim Investigational Site 353, Świętochłowice
  - Boehringer Ingelheim Investigational Site 359, Tarnobrzeg
  - Boehringer Ingelheim Investigational Site 362, Tarnowskie Góry
  - Boehringer Ingelheim Investigational Site 360, Tarnów
  - Boehringer Ingelheim Investigational Site 361, Tarnów
  - Boehringer Ingelheim Investigational Site 363, Tczew
  - Boehringer Ingelheim Investigational Site 364, Terespol
  - Boehringer Ingelheim Investigational Site 366, Tomaszow Maazowiecki
  - Boehringer Ingelheim Investigational Site 367, Tomaszow Maazowiecki
  - Boehringer Ingelheim Investigational Site 365, Tomaszów Lubelski
  - Boehringer Ingelheim Investigational Site 368, Torun
  - Boehringer Ingelheim Investigational Site 369, Torun
  - Boehringer Ingelheim Investigational Site 370, Torun
  - Boehringer Ingelheim Investigational Site 371, Torzym
  - Boehringer Ingelheim Investigational Site 372, Trzebnica
  - Boehringer Ingelheim Investigational Site 373, Twardogóra
  - Boehringer Ingelheim Investigational Site 374, Tychy
  - Boehringer Ingelheim Investigational Site 376, Urzedów
  - Boehringer Ingelheim Investigational Site 380, Warsaw
  - Boehringer Ingelheim Investigational Site 381, Warsaw
  - Boehringer Ingelheim Investigational Site 382, Warsaw
  - Boehringer Ingelheim Investigational Site 383, Warsaw
  - Boehringer Ingelheim Investigational Site 384, Warsaw
  - Boehringer Ingelheim Investigational Site 385, Warsaw
  - Boehringer Ingelheim Investigational Site 386, Warsaw
  - Boehringer Ingelheim Investigational Site 387, Warsaw
  - Boehringer Ingelheim Investigational Site 388, Warsaw
  - Boehringer Ingelheim Investigational Site 389, Warsaw
  - Boehringer Ingelheim Investigational Site 390, Warsaw
  - Boehringer Ingelheim Investigational Site 391, Warsaw
  - Boehringer Ingelheim Investigational Site 392, Warsaw
  - Boehringer Ingelheim Investigational Site 393, Warsaw
  - Boehringer Ingelheim Investigational Site 394, Warsaw
  - Boehringer Ingelheim Investigational Site 395, Warsaw
  - Boehringer Ingelheim Investigational Site 396, Warsaw
  - Boehringer Ingelheim Investigational Site 397, Warsaw
  - Boehringer Ingelheim Investigational Site 398, Warsaw
  - Boehringer Ingelheim Investigational Site 399, Warsaw
  - Boehringer Ingelheim Investigational Site 400, Warsaw
  - Boehringer Ingelheim Investigational Site 401, Warsaw
  - Boehringer Ingelheim Investigational Site 402, Warsaw
  - Boehringer Ingelheim Investigational Site 403, Warsaw
  - Boehringer Ingelheim Investigational Site 404, Warsaw
  - Boehringer Ingelheim Investigational Site 405, Warsaw
  - Boehringer Ingelheim Investigational Site 406, Warsaw
  - Boehringer Ingelheim Investigational Site 407, Warsaw
  - Boehringer Ingelheim Investigational Site 408, Warsaw
  - Boehringer Ingelheim Investigational Site 409, Warsaw
  - Boehringer Ingelheim Investigational Site 410, Warsaw
  - Boehringer Ingelheim Investigational Site 378, Wałbrzych
  - Boehringer Ingelheim Investigational Site 379, Wałcz
  - Boehringer Ingelheim Investigational Site 377, Wąbrzeźno
  - Boehringer Ingelheim Investigational Site 411, Wegrów
  - Boehringer Ingelheim Investigational Site 412, Wejherowo
  - Boehringer Ingelheim Investigational Site 413, Wejherowo
  - Boehringer Ingelheim Investigational Site 414, Wesoła
  - Boehringer Ingelheim Investigational Site 415, Wieliczka
  - Boehringer Ingelheim Investigational Site 416, Wieluń
  - Boehringer Ingelheim Investigational Site 417, Wieruszów
  - Boehringer Ingelheim Investigational Site 418, Wilkowice
  - Boehringer Ingelheim Investigational Site 419, Wilkowice
  - Boehringer Ingelheim Investigational Site 423, Wodzisław Śląski
  - Boehringer Ingelheim Investigational Site 424, Wojnicz
  - Boehringer Ingelheim Investigational Site 426, Wolsztyn
  - Boehringer Ingelheim Investigational Site 427, Wolsztyn
  - Boehringer Ingelheim Investigational Site 428, Wożniki
  - Boehringer Ingelheim Investigational Site 425, Wołomin
  - Boehringer Ingelheim Investigational Site 429, Wroclaw
  - Boehringer Ingelheim Investigational Site 430, Wroclaw
  - Boehringer Ingelheim Investigational Site 431, Wroclaw
  - Boehringer Ingelheim Investigational Site 432, Wroclaw
  - Boehringer Ingelheim Investigational Site 433, Wroclaw
  - Boehringer Ingelheim Investigational Site 434, Wroclaw
  - Boehringer Ingelheim Investigational Site 435, Września
  - Boehringer Ingelheim Investigational Site 436, Wyszków
  - Boehringer Ingelheim Investigational Site 420, Włocławek
  - Boehringer Ingelheim Investigational Site 421, Włocławek
  - Boehringer Ingelheim Investigational Site 422, Włocławek
  - Boehringer Ingelheim Investigational Site 438, Zabrze
  - Boehringer Ingelheim Investigational Site 439, Zabrze
  - Boehringer Ingelheim Investigational Site 440, Zabrze
  - Boehringer Ingelheim Investigational Site 441, Zakopane
  - Boehringer Ingelheim Investigational Site 442, Zambrów
  - Boehringer Ingelheim Investigational Site 443, Zamość
  - Boehringer Ingelheim Investigational Site 437, Ząbkowice Śląskie
  - Boehringer Ingelheim Investigational Site 445, Zblewo
  - Boehringer Ingelheim Investigational Site 446, Zduńska Wola
  - Boehringer Ingelheim Investigational Site 447, Zgierz
  - Boehringer Ingelheim Investigational Site 448, Zgierz
  - Boehringer Ingelheim Investigational Site 449, Zgorzelec
  - Boehringer Ingelheim Investigational Site 450, Zgorzelec
  - Boehringer Ingelheim Investigational Site 451, Zgorzelec
  - Boehringer Ingelheim Investigational Site 452, Zielona Góra
  - Boehringer Ingelheim Investigational Site 453, Zielona Góra
  - Boehringer Ingelheim Investigational Site 454, Zielonka
  - Boehringer Ingelheim Investigational Site 455, Zimnice Wielkie
  - Boehringer Ingelheim Investigational Site 456, Zlotów
  - Boehringer Ingelheim Investigational Site 458, Zyradow
  - Boehringer Ingelheim Investigational Site 459, Zyradow
  - Boehringer Ingelheim Investigational Site 444, Żary
  - Boehringer Ingelheim Investigational Site 457, Żnin
  - Boehringer Ingelheim Investigational Site 460, Żywiec
  - Boehringer Ingelheim Investigational Site 180, Łańcut
  - Boehringer Ingelheim Investigational Site 201, Łomża
- Romania (86):
  - Boehringer Ingelheim Investigational Site 461, Arad
  - Boehringer Ingelheim Investigational Site 462, Bacau
  - Boehringer Ingelheim Investigational Site 463, Bacau
  - Boehringer Ingelheim Investigational Site 464, Bacau
  - Boehringer Ingelheim Investigational Site 465, Baia Mare
  - Boehringer Ingelheim Investigational Site 466, Bârlad
  - Boehringer Ingelheim Investigational Site 467, Botoșani
  - Boehringer Ingelheim Investigational Site 469, Brasov
  - Boehringer Ingelheim Investigational Site 470, Brasov
  - Boehringer Ingelheim Investigational Site 468, Brăila
  - Boehringer Ingelheim Investigational Site 471, Breaza
  - Boehringer Ingelheim Investigational Site 472, Bucharest
  - Boehringer Ingelheim Investigational Site 473, Bucharest
  - Boehringer Ingelheim Investigational Site 474, Bucharest
  - Boehringer Ingelheim Investigational Site 475, Bucharest
  - Boehringer Ingelheim Investigational Site 476, Bucharest
  - Boehringer Ingelheim Investigational Site 477, Bucharest
  - Boehringer Ingelheim Investigational Site 478, Bucharest
  - Boehringer Ingelheim Investigational Site 479, Bucharest
  - Boehringer Ingelheim Investigational Site 480, Bucharest
  - Boehringer Ingelheim Investigational Site 481, Bucharest
  - Boehringer Ingelheim Investigational Site 482, Bucharest
  - Boehringer Ingelheim Investigational Site 483, Bucharest
  - Boehringer Ingelheim Investigational Site 484, Bucharest
  - Boehringer Ingelheim Investigational Site 485, Buzău
  - Boehringer Ingelheim Investigational Site 486, Buzău
  - Boehringer Ingelheim Investigational Site 488, Campulung Muscel
  - Boehringer Ingelheim Investigational Site 487, Câmpina
  - Boehringer Ingelheim Investigational Site 489, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 490, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 491, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 492, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 493, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 494, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 495, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 496, Constanța
  - Boehringer Ingelheim Investigational Site 497, Constanța
  - Boehringer Ingelheim Investigational Site 498, Constanța
  - Boehringer Ingelheim Investigational Site 499, Constanța
  - Boehringer Ingelheim Investigational Site 500, Craiova
  - Boehringer Ingelheim Investigational Site 501, Craiova
  - Boehringer Ingelheim Investigational Site 502, Craiova
  - Boehringer Ingelheim Investigational Site 503, Deva
  - Boehringer Ingelheim Investigational Site 504, Drajna de Jos
  - Boehringer Ingelheim Investigational Site 505, Drobeta-Turnu Severin
  - Boehringer Ingelheim Investigational Site 506, Galati
  - Boehringer Ingelheim Investigational Site 507, Galati
  - Boehringer Ingelheim Investigational Site 508, Galati
  - Boehringer Ingelheim Investigational Site 509, Galati
  - Boehringer Ingelheim Investigational Site 510, Galati
  - Boehringer Ingelheim Investigational Site 511, Giurgiu
  - Boehringer Ingelheim Investigational Site 512, Hunedoara
  - Boehringer Ingelheim Investigational Site 513, Iași
  - Boehringer Ingelheim Investigational Site 514, Iași
  - Boehringer Ingelheim Investigational Site 515, Iași
  - Boehringer Ingelheim Investigational Site 516, Iași
  - Boehringer Ingelheim Investigational Site 517, Leordeni
  - Boehringer Ingelheim Investigational Site 518, Marghita
  - Boehringer Ingelheim Investigational Site 519, Mures
  - Boehringer Ingelheim Investigational Site 520, Mures
  - Boehringer Ingelheim Investigational Site 521, Mures
  - Boehringer Ingelheim Investigational Site 522, Neamt
  - Boehringer Ingelheim Investigational Site 523, Onești
  - Boehringer Ingelheim Investigational Site 524, Oradea
  - Boehringer Ingelheim Investigational Site 525, Oradea
  - Boehringer Ingelheim Investigational Site 526, Oradea
  - Boehringer Ingelheim Investigational Site 527, Piteşti
  - Boehringer Ingelheim Investigational Site 528, Piteşti
  - Boehringer Ingelheim Investigational Site 529, Ploieşti
  - Boehringer Ingelheim Investigational Site 530, Ploieşti
  - Boehringer Ingelheim Investigational Site 531, Ploieşti
  - Boehringer Ingelheim Investigational Site 532, Râmnicu Vâlcea
  - Boehringer Ingelheim Investigational Site 533, Râmnicu Vâlcea
  - Boehringer Ingelheim Investigational Site 534, Roșiorii de Vede
  - Boehringer Ingelheim Investigational Site 535, Satu Mare
  - Boehringer Ingelheim Investigational Site 536, Scorniceşti
  - Boehringer Ingelheim Investigational Site 537, Scorniceşti
  - Boehringer Ingelheim Investigational Site 538, Suceava
  - Boehringer Ingelheim Investigational Site 539, Suceava
  - Boehringer Ingelheim Investigational Site 540, Suceava
  - Boehringer Ingelheim Investigational Site 541, Târgovişte
  - Boehringer Ingelheim Investigational Site 542, Târgovişte
  - Boehringer Ingelheim Investigational Site 543, Timișoara
  - Boehringer Ingelheim Investigational Site 544, Timișoara
  - Boehringer Ingelheim Investigational Site 545, Timișoara
  - Boehringer Ingelheim Investigational Site 546, Zalău
- Russia (188):
  - Boehringer Ingelheim Investigational Site 547, Astrakhan
  - Boehringer Ingelheim Investigational Site 548, Astrakhan
  - Boehringer Ingelheim Investigational Site 549, Barnaul
  - Boehringer Ingelheim Investigational Site 550, Belgorod
  - Boehringer Ingelheim Investigational Site 551, Chelyabinsk
  - Boehringer Ingelheim Investigational Site 552, Chelyabinsk
  - Boehringer Ingelheim Investigational Site 553, Chelyabinsk
  - Boehringer Ingelheim Investigational Site 554, Dinskaya
  - Boehringer Ingelheim Investigational Site 555, Engel's
  - Boehringer Ingelheim Investigational Site 561, Gatchina
  - Boehringer Ingelheim Investigational Site 562, Izhevsk
  - Boehringer Ingelheim Investigational Site 563, Izhevsk
  - Boehringer Ingelheim Investigational Site 564, Kaluga
  - Boehringer Ingelheim Investigational Site 565, Kaluga
  - Boehringer Ingelheim Investigational Site 566, Kaluga
  - Boehringer Ingelheim Investigational Site 567, Kazan'
  - Boehringer Ingelheim Investigational Site 568, Kazan'
  - Boehringer Ingelheim Investigational Site 569, Kazan'
  - Boehringer Ingelheim Investigational Site 570, Kazan'
  - Boehringer Ingelheim Investigational Site 571, Kazan'
  - Boehringer Ingelheim Investigational Site 572, Kemerovo
  - Boehringer Ingelheim Investigational Site 573, Kemerovo
  - Boehringer Ingelheim Investigational Site 574, Kemerovo
  - Boehringer Ingelheim Investigational Site 575, Kemerovo
  - Boehringer Ingelheim Investigational Site 576, Kemerovo
  - Boehringer Ingelheim Investigational Site 577, Khabarovsk
  - Boehringer Ingelheim Investigational Site 578, Khabarovsk
  - Boehringer Ingelheim Investigational Site 579, Kirov
  - Boehringer Ingelheim Investigational Site 580, Klintsy of Bryansk Region
  - Boehringer Ingelheim Investigational Site 581, Korolyov
  - Boehringer Ingelheim Investigational Site 582, Krasnodar
  - Boehringer Ingelheim Investigational Site 583, Krasnodar
  - Boehringer Ingelheim Investigational Site 584, Krasnodar
  - Boehringer Ingelheim Investigational Site 585, Krasnodar
  - Boehringer Ingelheim Investigational Site 586, Krasnoyarsk
  - Boehringer Ingelheim Investigational Site 587, Krasnoyarsk
  - Boehringer Ingelheim Investigational Site 588, Krasnoyarsk
  - Boehringer Ingelheim Investigational Site 589, Krasnoyarsk
  - Boehringer Ingelheim Investigational Site 590, Krasnoyarsk
  - Boehringer Ingelheim Investigational Site 591, Krasnoyarsk
  - Boehringer Ingelheim Investigational Site 592, Kursk
  - Boehringer Ingelheim Investigational Site 593, Lipetsk
  - Boehringer Ingelheim Investigational Site 594, Magnitogorsk
  - Boehringer Ingelheim Investigational Site 595, Makhachkala
  - Boehringer Ingelheim Investigational Site 596, Mine
  - Boehringer Ingelheim Investigational Site 597, Moscow
  - Boehringer Ingelheim Investigational Site 598, Moscow
  - Boehringer Ingelheim Investigational Site 599, Moscow
  - Boehringer Ingelheim Investigational Site 600, Moscow
  - Boehringer Ingelheim Investigational Site 601, Moscow
  - Boehringer Ingelheim Investigational Site 602, Moscow
  - Boehringer Ingelheim Investigational Site 603, Moscow
  - Boehringer Ingelheim Investigational Site 604, Moscow
  - Boehringer Ingelheim Investigational Site 605, Moscow
  - Boehringer Ingelheim Investigational Site 606, Moscow
  - Boehringer Ingelheim Investigational Site 607, Moscow
  - Boehringer Ingelheim Investigational Site 608, Moscow
  - Boehringer Ingelheim Investigational Site 609, Moscow
  - Boehringer Ingelheim Investigational Site 610, Moscow
  - Boehringer Ingelheim Investigational Site 611, Moscow
  - Boehringer Ingelheim Investigational Site 612, Moscow
  - Boehringer Ingelheim Investigational Site 613, Moscow
  - Boehringer Ingelheim Investigational Site 614, Moscow
  - Boehringer Ingelheim Investigational Site 615, Moscow
  - Boehringer Ingelheim Investigational Site 616, Moscow
  - Boehringer Ingelheim Investigational Site 617, Moscow
  - Boehringer Ingelheim Investigational Site 618, Moscow
  - Boehringer Ingelheim Investigational Site 619, Moscow
  - Boehringer Ingelheim Investigational Site 620, Moscow
  - Boehringer Ingelheim Investigational Site 621, Moscow
  - Boehringer Ingelheim Investigational Site 622, Moscow
  - Boehringer Ingelheim Investigational Site 623, Moscow
  - Boehringer Ingelheim Investigational Site 624, Moscow
  - Boehringer Ingelheim Investigational Site 625, Moscow
  - Boehringer Ingelheim Investigational Site 626, Moscow
  - Boehringer Ingelheim Investigational Site 627, Moscow
  - Boehringer Ingelheim Investigational Site 628, Moscow
  - Boehringer Ingelheim Investigational Site 629, Moscow
  - Boehringer Ingelheim Investigational Site 630, Moscow
  - Boehringer Ingelheim Investigational Site 631, Moscow
  - Boehringer Ingelheim Investigational Site 632, Moscow
  - Boehringer Ingelheim Investigational Site 633, Moscow
  - Boehringer Ingelheim Investigational Site 634, Moscow
  - Boehringer Ingelheim Investigational Site 635, Moscow
  - Boehringer Ingelheim Investigational Site 636, Moscow
  - Boehringer Ingelheim Investigational Site 637, Moscow
  - Boehringer Ingelheim Investigational Site 638, Moscow
  - Boehringer Ingelheim Investigational Site 639, Moscow
  - Boehringer Ingelheim Investigational Site 640, Moscow
  - Boehringer Ingelheim Investigational Site 642, Nal'chik
  - Boehringer Ingelheim Investigational Site 643, Naro-Fominsk
  - Boehringer Ingelheim Investigational Site 644, Nefteugansk
  - Boehringer Ingelheim Investigational Site 641, Nizhny Novgorod
  - Boehringer Ingelheim Investigational Site 645, Nizhny Tagil
  - Boehringer Ingelheim Investigational Site 646, Nizhny Tagil
  - Boehringer Ingelheim Investigational Site 647, Noginsk
  - Boehringer Ingelheim Investigational Site 648, Novokuznetsk
  - Boehringer Ingelheim Investigational Site 649, Novokuznetsk
  - Boehringer Ingelheim Investigational Site 650, Novokuznetsk
  - Boehringer Ingelheim Investigational Site 651, Novosibirsk
  - Boehringer Ingelheim Investigational Site 652, Novosibirsk
  - Boehringer Ingelheim Investigational Site 653, Novosibirsk
  - Boehringer Ingelheim Investigational Site 654, Odintsovo
  - Boehringer Ingelheim Investigational Site 655, Omsk
  - Boehringer Ingelheim Investigational Site 656, Orenburg
  - Boehringer Ingelheim Investigational Site 657, Orenburg
  - Boehringer Ingelheim Investigational Site 658, Penza
  - Boehringer Ingelheim Investigational Site 659, Penza
  - Boehringer Ingelheim Investigational Site 660, Perm
  - Boehringer Ingelheim Investigational Site 661, Perm
  - Boehringer Ingelheim Investigational Site 662, Perm
  - Boehringer Ingelheim Investigational Site 663, Pushkino
  - Boehringer Ingelheim Investigational Site 664, Pyatigorsk
  - Boehringer Ingelheim Investigational Site 665, Ramenskoye
  - Boehringer Ingelheim Investigational Site 666, Rostov-on-Donu
  - Boehringer Ingelheim Investigational Site 667, Rostov-on-Donu
  - Boehringer Ingelheim Investigational Site 668, Rostov-on-Donu
  - Boehringer Ingelheim Investigational Site 669, Rostov-on-Donu
  - Boehringer Ingelheim Investigational Site 670, Ryazan
  - Boehringer Ingelheim Investigational Site 671, Ryazan
  - Boehringer Ingelheim Investigational Site 672, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 673, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 674, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 675, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 676, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 677, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 678, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 679, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 680, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 681, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 682, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 683, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 684, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 685, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 686, Samara
  - Boehringer Ingelheim Investigational Site 687, Samara
  - Boehringer Ingelheim Investigational Site 688, Saratov
  - Boehringer Ingelheim Investigational Site 689, Saratov
  - Boehringer Ingelheim Investigational Site 690, Saratov
  - Boehringer Ingelheim Investigational Site 691, Saratov
  - Boehringer Ingelheim Investigational Site 692, Saratov
  - Boehringer Ingelheim Investigational Site 693, Saratov
  - Boehringer Ingelheim Investigational Site 694, Saratov
  - Boehringer Ingelheim Investigational Site 695, Smolensk
  - Boehringer Ingelheim Investigational Site 696, Sochi
  - Boehringer Ingelheim Investigational Site 697, Stavropol
  - Boehringer Ingelheim Investigational Site 698, Stavropol
  - Boehringer Ingelheim Investigational Site 699, Stavropol
  - Boehringer Ingelheim Investigational Site 700, Surgut
  - Boehringer Ingelheim Investigational Site 701, Taganrog
  - Boehringer Ingelheim Investigational Site 702, Tolyatti
  - Boehringer Ingelheim Investigational Site 703, Tolyatti
  - Boehringer Ingelheim Investigational Site 704, Tolyatti
  - Boehringer Ingelheim Investigational Site 705, Tomsk
  - Boehringer Ingelheim Investigational Site 706, Tomsk
  - Boehringer Ingelheim Investigational Site 707, Tomsk
  - Boehringer Ingelheim Investigational Site 708, Tomsk
  - Boehringer Ingelheim Investigational Site 709, Tula
  - Boehringer Ingelheim Investigational Site 712, Tver'
  - Boehringer Ingelheim Investigational Site 710, Tyumen
  - Boehringer Ingelheim Investigational Site 711, Tyumen
  - Boehringer Ingelheim Investigational Site 713, Ufa
  - Boehringer Ingelheim Investigational Site 714, Ufa
  - Boehringer Ingelheim Investigational Site 715, Ufa
  - Boehringer Ingelheim Investigational Site 716, Ufa
  - Boehringer Ingelheim Investigational Site 717, Ufa
  - Boehringer Ingelheim Investigational Site 718, Ufa
  - Boehringer Ingelheim Investigational Site 719, Ulan-Ude
  - Boehringer Ingelheim Investigational Site 720, Ulan-Ude
  - Boehringer Ingelheim Investigational Site 721, Ulyanovsk
  - Boehringer Ingelheim Investigational Site 722, Ulyanovsk
  - Boehringer Ingelheim Investigational Site 723, Vladikavkaz
  - Boehringer Ingelheim Investigational Site 724, Vladimir
  - Boehringer Ingelheim Investigational Site 725, Vladimir
  - Boehringer Ingelheim Investigational Site 726, Volgograd
  - Boehringer Ingelheim Investigational Site 727, Volgograd
  - Boehringer Ingelheim Investigational Site 728, Volgograd
  - Boehringer Ingelheim Investigational Site 729, Voronezh
  - Boehringer Ingelheim Investigational Site 730, Voronezh
  - Boehringer Ingelheim Investigational Site 731, Voronezh
  - Boehringer Ingelheim Investigational Site 732, Yaroslavl
  - Boehringer Ingelheim Investigational Site 556, Yekaterinburg
  - Boehringer Ingelheim Investigational Site 557, Yekaterinburg
  - Boehringer Ingelheim Investigational Site 558, Yekaterinburg
  - Boehringer Ingelheim Investigational Site 559, Yekaterinburg
  - Boehringer Ingelheim Investigational Site 560, Yekaterinburg
  - Boehringer Ingelheim Investigational Site 733, Zheleznogorsk
  - Boehringer Ingelheim Investigational Site 734, Zheleznogorsk
- Slovakia (93):
  - Boehringer Ingelheim Investigational Site 735, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 736, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 737, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 738, Bardejov
  - Boehringer Ingelheim Investigational Site 739, Bardejov
  - Boehringer Ingelheim Investigational Site 740, Bojnice
  - Boehringer Ingelheim Investigational Site 741, Bratislava
  - Boehringer Ingelheim Investigational Site 742, Bratislava
  - Boehringer Ingelheim Investigational Site 743, Bratislava
  - Boehringer Ingelheim Investigational Site 744, Bratislava
  - Boehringer Ingelheim Investigational Site 745, Bratislava
  - Boehringer Ingelheim Investigational Site 746, Bratislava
  - Boehringer Ingelheim Investigational Site 747, Bratislava
  - Boehringer Ingelheim Investigational Site 748, Bratislava
  - Boehringer Ingelheim Investigational Site 749, Brezno
  - Boehringer Ingelheim Investigational Site 750, Brezno
  - Boehringer Ingelheim Investigational Site 751, Čadca
  - Boehringer Ingelheim Investigational Site 752, Galanta
  - Boehringer Ingelheim Investigational Site 753, Hurbanovo
  - Boehringer Ingelheim Investigational Site 754, Ilava
  - Boehringer Ingelheim Investigational Site 755, Kežmarok
  - Boehringer Ingelheim Investigational Site 756, Košice
  - Boehringer Ingelheim Investigational Site 757, Košice
  - Boehringer Ingelheim Investigational Site 758, Košice
  - Boehringer Ingelheim Investigational Site 759, Košice
  - Boehringer Ingelheim Investigational Site 760, Košice
  - Boehringer Ingelheim Investigational Site 761, Košice
  - Boehringer Ingelheim Investigational Site 762, Košice
  - Boehringer Ingelheim Investigational Site 763, Krompachy
  - Boehringer Ingelheim Investigational Site 764, Kysúcke Nové Mesto
  - Boehringer Ingelheim Investigational Site 765, Levice
  - Boehringer Ingelheim Investigational Site 766, Levoča
  - Boehringer Ingelheim Investigational Site 767, Liptovský Hrádok
  - Boehringer Ingelheim Investigational Site 768, Lučenec
  - Boehringer Ingelheim Investigational Site 769, Lučenec
  - Boehringer Ingelheim Investigational Site 770, Lučenec
  - Boehringer Ingelheim Investigational Site 771, Malacky
  - Boehringer Ingelheim Investigational Site 772, Martin
  - Boehringer Ingelheim Investigational Site 773, Martin
  - Boehringer Ingelheim Investigational Site 774, Medzilaborce
  - Boehringer Ingelheim Investigational Site 775, Michalovce
  - Boehringer Ingelheim Investigational Site 776, Michalovce
  - Boehringer Ingelheim Investigational Site 777, Michalovce
  - Boehringer Ingelheim Investigational Site 778, Moldava nad Bodvou
  - Boehringer Ingelheim Investigational Site 779, Myjava
  - Boehringer Ingelheim Investigational Site 780, Nitra
  - Boehringer Ingelheim Investigational Site 781, Nitra
  - Boehringer Ingelheim Investigational Site 782, Nitra
  - Boehringer Ingelheim Investigational Site 783, Nová Bana
  - Boehringer Ingelheim Investigational Site 784, Nováky
  - Boehringer Ingelheim Investigational Site 785, Nové Mesto nad Váhom
  - Boehringer Ingelheim Investigational Site 786, Nové Mesto nad Váhom
  - Boehringer Ingelheim Investigational Site 787, Nové Zámky
  - Boehringer Ingelheim Investigational Site 788, Nové Zámky
  - Boehringer Ingelheim Investigational Site 789, Nové Zámky
  - Boehringer Ingelheim Investigational Site 790, Poprad
  - Boehringer Ingelheim Investigational Site 791, Povazská Bystrica
  - Boehringer Ingelheim Investigational Site 792, Prešov
  - Boehringer Ingelheim Investigational Site 793, Prešov
  - Boehringer Ingelheim Investigational Site 794, Prievidza
  - Boehringer Ingelheim Investigational Site 795, Prievidza
  - Boehringer Ingelheim Investigational Site 796, Rimavská Sobota
  - Boehringer Ingelheim Investigational Site 797, Rimavská Sobota
  - Boehringer Ingelheim Investigational Site 798, Rožňava
  - Boehringer Ingelheim Investigational Site 799, Rožňava
  - Boehringer Ingelheim Investigational Site 801, Senec
  - Boehringer Ingelheim Investigational Site 802, Sereď
  - Boehringer Ingelheim Investigational Site 803, Skalica
  - Boehringer Ingelheim Investigational Site 804, Snina
  - Boehringer Ingelheim Investigational Site 805, Sp. Nová Ves
  - Boehringer Ingelheim Investigational Site 806, Sp. Nová Ves
  - Boehringer Ingelheim Investigational Site 807, Stará Lubovna
  - Boehringer Ingelheim Investigational Site 808, Stropkov
  - Boehringer Ingelheim Investigational Site 809, Stúrovo
  - Boehringer Ingelheim Investigational Site 811, Svidník
  - Boehringer Ingelheim Investigational Site 800, Šamorín
  - Boehringer Ingelheim Investigational Site 810, Šurany
  - Boehringer Ingelheim Investigational Site 812, Topoľčany
  - Boehringer Ingelheim Investigational Site 813, Trebišov
  - Boehringer Ingelheim Investigational Site 814, Trenčín
  - Boehringer Ingelheim Investigational Site 815, Trnava
  - Boehringer Ingelheim Investigational Site 816, Trnava
  - Boehringer Ingelheim Investigational Site 817, Trstená
  - Boehringer Ingelheim Investigational Site 818, Velké Kapusany
  - Boehringer Ingelheim Investigational Site 819, Velký Krtis
  - Boehringer Ingelheim Investigational Site 821, Vranov n/Toplou
  - Boehringer Ingelheim Investigational Site 822, Vranov n/Toplou
  - Boehringer Ingelheim Investigational Site 820, Vráble
  - Boehringer Ingelheim Investigational Site 825, Zvolen
  - Boehringer Ingelheim Investigational Site 826, Zvolen
  - Boehringer Ingelheim Investigational Site 827, Zvolen
  - Boehringer Ingelheim Investigational Site 823, Žiar nad Hronom
  - Boehringer Ingelheim Investigational Site 824, Žilina
- Slovenia (37):
  - Boehringer Ingelheim Investigational Site 828, Celje
  - Boehringer Ingelheim Investigational Site 829, Celje
  - Boehringer Ingelheim Investigational Site 830, Celje
  - Boehringer Ingelheim Investigational Site 831, Celje
  - Boehringer Ingelheim Investigational Site 832, Celje
  - Boehringer Ingelheim Investigational Site 833, Domžale
  - Boehringer Ingelheim Investigational Site 834, Golnik
  - Boehringer Ingelheim Investigational Site 835, Grosuplje
  - Boehringer Ingelheim Investigational Site 836, Jesenice
  - Boehringer Ingelheim Investigational Site 837, Kamnik
  - Boehringer Ingelheim Investigational Site 838, Kočevje
  - Boehringer Ingelheim Investigational Site 839, Koper
  - Boehringer Ingelheim Investigational Site 840, Kranj
  - Boehringer Ingelheim Investigational Site 841, Kranj
  - Boehringer Ingelheim Investigational Site 842, Litija
  - Boehringer Ingelheim Investigational Site 843, Ljubljana
  - Boehringer Ingelheim Investigational Site 844, Ljubljana
  - Boehringer Ingelheim Investigational Site 845, Ljubljana
  - Boehringer Ingelheim Investigational Site 846, Ljubljana
  - Boehringer Ingelheim Investigational Site 847, Maribor
  - Boehringer Ingelheim Investigational Site 848, Maribor
  - Boehringer Ingelheim Investigational Site 849, Maribor
  - Boehringer Ingelheim Investigational Site 850, Murska Sobota
  - Boehringer Ingelheim Investigational Site 851, Murska Sobota
  - Boehringer Ingelheim Investigational Site 852, Murska Sobota
  - Boehringer Ingelheim Investigational Site 853, Nova Gorica
  - Boehringer Ingelheim Investigational Site 854, Portorož
  - Boehringer Ingelheim Investigational Site 855, Ptuj
  - Boehringer Ingelheim Investigational Site 856, Ptuj
  - Boehringer Ingelheim Investigational Site 857, Radovljica
  - Boehringer Ingelheim Investigational Site 858, Ravne na Koroškem
  - Boehringer Ingelheim Investigational Site 859, Sežana
  - Boehringer Ingelheim Investigational Site 860, Sežana
  - Boehringer Ingelheim Investigational Site 861, Slovenj Gradec
  - Boehringer Ingelheim Investigational Site 862, Slovenska Bistrica
  - Boehringer Ingelheim Investigational Site 863, Velenje
  - Boehringer Ingelheim Investigational Site 864, Vrhnika

REFERENCES:
- [Derived] Flezar M, Jahnz-Rozyk K, Enache G, Martynenko T, Kristufek P, Skrinjaric-Cincar S, Kadlecova P, Martinovic G. SOSPES: SPIRIVA(R) observational study measuring SGRQ score in routine medical practice in Central and Eastern Europe. Int J Chron Obstruct Pulmon Dis. 2013;8:483-92. doi: 10.2147/COPD.S45640. Epub 2013 Oct 9. PMID 24159258

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Whilst 4854 patients were enrolled in the study, only 4852 of these entered and were included in the treated set, since two patients had no evidence of Spiriva administration.
Groups:
- Patients Treated With Spiriva: Treatment with 18 mcg tiotropium inhalation capsules of Spiriva
Period: Overall Study
Arm/Group | Patients Treated With Spiriva
Started | 4852
Completed | 4712
Not Completed | 140
Not completed — Adverse Event | 22
Not completed — Protocol Violation | 14
Not completed — Lost to Follow-up | 32
Not completed — Other | 72

BASELINE CHARACTERISTICS:
Arm/Group | Patients Treated With Spiriva
Number analyzed (Participants) | 4852
Age, Continuous [Mean (Standard Deviation); unit: Years] — There were only 4779 patients with a non-missing age.
  Years | 62.6 (9.8)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 3433
  Female | 1391
  Missing | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of Total Saint George Respiratory Questionnaire (SGRQ) Score at the End of the Observational Period After 6 Months From Baseline
Description: The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life)
Time Frame: Baseline and 6 months
Population: Patients from the treated set (TS) who have evaluable SGRQ measurements at baseline and Visit 3 (6 months)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients Treated With Spiriva
Number analyzed (Participants) | 4335
Units on a scale | -21.73 (19.09)

2. Secondary Outcome: Additional Bronchodilator or Inhaled Corticosteroids (ICS)
Description: Pulmonary medication from baseline to visit 3 (6 months)
Time Frame: 6 months
Population: Patients from Full Analysis Set (FAS) which includes all patients from the TS who were assessed after administration of Spiriva, i.e. who have evaluable SGRQ measurements at visit 2 or visit 3.
Measure: Number; unit: Number of participants
Arm/Group | Patients Treated With Spiriva
Number analyzed (Participants) | 4435
Number of participants | 1146

3. Secondary Outcome: Compliance of Patients
Description: Patients are considered to be compliant if the difference of the number of days between visit 1 (baseline) and visit 3 (6months) and the number of actual taken capsules is less than 10.
Time Frame: 6 months
Population: Patients from FAS
Measure: Number; unit: Number of participants
Arm/Group | Patients Treated With Spiriva
Number analyzed (Participants) | 4435
Number of participants | 3636

4. Secondary Outcome: Patients With Any Adverse Events
Time Frame: 6 months
Population: TS
Measure: Number; unit: Number of participants
Arm/Group | Patients Treated With Spiriva
Number analyzed (Participants) | 4852
Number of participants | 182

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients Treated With Spiriva
Serious Adverse Events (participants affected / at risk) | 15/4852
Other Adverse Events (participants affected / at risk) | 0/4852
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With Spiriva (N=4852)
Brain oedema (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Tongue neoplasm malignant stage unspecified (Gastrointestinal disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Death (General disorders) | 1
Pyrexia (General disorders) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.